CLINICAL TRIAL: NCT00987129
Title: Effect of Omega-6:Omega-3 Fatty Acid Ratio on Delaying Progression of Age-related Macular Degeneration (AMD) in Moderate to High Risk Individuals.
Brief Title: Omega 6:Omega 3 Ratio and Progression of Age-related Macular Degeneration (AMD).
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: Yves Sauve (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Yves Sauve, PhD, AHFMR Senior Scholar, Ophthalmology Assistant Professor, University of Alberta, University of Alberta
Organization: University of Alberta (Other)
Other Study IDs: MOP 79278; 200809MOP-192321; CIA-CBAA-27683
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2012-08

CONDITIONS: Age-related Macular Degeneration
Keywords: DHA; EPA; AMD; drusen; omega-3 fatty acids; omega6:omega3 ratio
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for genotyping and measuring omega-3 FA status. Serum for Cytokine level analysis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Docosahexaenoic acid (DHA) supplementation has been shown to prevent specific age-related changes in the retina through biochemical and functional evaluations, but it is unclear whether increased DHA intake-reflected through elevated DHA+EPA blood levels-can affect the natural history and progression of age-related macular degeneration (AMD). AMD is a disease affecting the macula, the part of the eye containing cone photoreceptors at the center of the visual field. The macula is responsible for vision in most daily functions, including reading, seeing fine details, and colour recognition. Severe AMD can lead to a central scotoma, severely impairing daily functioning. AMD can be divided into two forms: the more severe wet AMD, consisting of proliferation of new blood vessels in the retina, and dry AMD characterized by the development of drusen, a buildup of extracellular material . The investigators are focused on the group with the highest risk of developing the two advanced forms of AMD [wet AMD or central geographic atrophy]: patients with unilateral wet AMD and dry AMD in their other eye. The study will consist of following up a cohort of such subjects and monitoring their visual function in a comprehensive manner. Working in concert with clinical ophthalmologists and basic scientists, the investigators will monitor "DHA+EPA" and "Omega6:Omega3 fatty acid ratio" levels in the blood, inherited predispositions through genetic analysis, lipofuscin (an accumulated waste product) levels & AMD progression via fundus photography, visual acuity, and retinal function via full-field and multifocal electroretinograms. These different factors will be cross-correlated and evaluated to determine how omega-3 fatty acids affect the progression of AMD.

ELIGIBILITY:
Inclusion Criteria:

* 50+ years of age
* NVAMD (Wet) in one eye, early or intermediate dry-AMD in the fellow eye
* taking AREDS vitamins (or equivalent)

Exclusion Criteria:

* Central geographic atrophy
* Diabetic retinopathy
* Ocular surgery in the eye with dry-AMD (not including cataract IOL surgery)
* Underlying ocular pathology in the eye with dry-AMD (especially glaucoma, dense cataracts, and retinitis pigmentosa)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with Neovascular (wet) AMD in one eye and early or intermediate dry AMD in the fellow eye, taking AREDS vitamins (or equivalent).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Progression of dry AMD status according to international classification/grading system. | 2 year

SECONDARY OUTCOMES:
Delayed progression to neovascular AMD (NVAMD) or Central Geographic Atrophy (cGA) in the fellow eye. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yves Sauvé, PhD, Principal Investigator — Department of Ophthalmology
Locations (3):
- Canada (3):
  - Alberta Retina Consultants, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta

REFERENCES:
- [Background] Chiu CJ, Klein R, Milton RC, Gensler G, Taylor A. Does eating particular diets alter the risk of age-related macular degeneration in users of the Age-Related Eye Disease Study supplements? Br J Ophthalmol. 2009 Sep;93(9):1241-6. doi: 10.1136/bjo.2008.143412. Epub 2009 Jun 9. PMID 19508997
- [Background] Cakiner-Egilmez T. Omega 3 fatty acids and the eye. Insight. 2008 Oct-Dec;33(4):20-5; quiz 26-7. PMID 19227095
- [Background] Querques G, Benlian P, Chanu B, Portal C, Coscas G, Soubrane G, Souied EH. Nutritional AMD treatment phase I (NAT-1): feasibility of oral DHA supplementation in age-related macular degeneration. Eur J Ophthalmol. 2009 Jan-Feb;19(1):100-6. doi: 10.1177/112067210901900115. PMID 19123156
- [Background] SanGiovanni JP, Chew EY, Agron E, Clemons TE, Ferris FL 3rd, Gensler G, Lindblad AS, Milton RC, Seddon JM, Klein R, Sperduto RD; Age-Related Eye Disease Study Research Group. The relationship of dietary omega-3 long-chain polyunsaturated fatty acid intake with incident age-related macular degeneration: AREDS report no. 23. Arch Ophthalmol. 2008 Sep;126(9):1274-9. doi: 10.1001/archopht.126.9.1274. PMID 18779490
- [Background] Augood C, Chakravarthy U, Young I, Vioque J, de Jong PT, Bentham G, Rahu M, Seland J, Soubrane G, Tomazzoli L, Topouzis F, Vingerling JR, Fletcher AE. Oily fish consumption, dietary docosahexaenoic acid and eicosapentaenoic acid intakes, and associations with neovascular age-related macular degeneration. Am J Clin Nutr. 2008 Aug;88(2):398-406. doi: 10.1093/ajcn/88.2.398. PMID 18689376
- [Background] Johnson EJ, Chung HY, Caldarella SM, Snodderly DM. The influence of supplemental lutein and docosahexaenoic acid on serum, lipoproteins, and macular pigmentation. Am J Clin Nutr. 2008 May;87(5):1521-9. doi: 10.1093/ajcn/87.5.1521. PMID 18469279
- [Background] Huang LL, Coleman HR, Kim J, de Monasterio F, Wong WT, Schleicher RL, Ferris FL 3rd, Chew EY. Oral supplementation of lutein/zeaxanthin and omega-3 long chain polyunsaturated fatty acids in persons aged 60 years or older, with or without AMD. Invest Ophthalmol Vis Sci. 2008 Sep;49(9):3864-9. doi: 10.1167/iovs.07-1420. Epub 2008 Apr 30. PMID 18450596